CLINICAL TRIAL: NCT07394881
Title: Do Video Animations and 3-D Skull Models Reduce Preoperative Anxiety in Bimaxillary Orthognathic Surgery Patients? Single Blinded Randomized Controlled Trial
Brief Title: Visual Tools and Preoperative Anxiety in Orthognathic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Uğur Boz, Oral and Maxillofacial Surgery Resident, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24/159
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Preoperative Anxiety; Orthognathic Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Three-arm, parallel-group randomized study comparing standard counseling alone versus counseling supplemented with a video animation or a 3-D skull model.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments were administered by blinded personnel who were not involved in delivering the information sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Standardized verbal preoperative information.
  Interventions: Behavioral: Verbal İnformation
- Video Animation Tools (Experimental): animation video used as a visual tool during counseling.
  Interventions: Behavioral: Animation Video Counseling
- 3D-Head Skull Tools (Experimental): Anatomical skull model demonstration used as a visual tool during counseling.
  Interventions: Behavioral: 3-D Skull Model Counseling

INTERVENTIONS:
Behavioral: Verbal İnformation — Standardized preoperative verbal information provided to all participants.
  Arms: Control
Behavioral: Animation Video Counseling — Standardized preoperative verbal counseling supplemented with an animation video explaining the surgical procedure and potential complications.
  Arms: Video Animation Tools
Behavioral: 3-D Skull Model Counseling — Standardized preoperative verbal counseling supplemented with a 3-D anatomical skull model demonstration to explain surgical anatomy and the planned procedure.
  Arms: 3D-Head Skull Tools

SUMMARY:
This study evaluates whether adding visual tools to standard preoperative counseling can reduce anxiety in patients scheduled for bimaxillary orthognathic surgery. Participants aged 18-36 years undergoing elective surgery was randomly assigned to one of three groups: (1) standard verbal information, (2) standard verbal information with a short animation video, (3) standard verbal information with a 3-D anatomical skull model demonstration. Anxiety was assessed using the State-Trait Anxiety Inventory and a visual analog scale at two time points: before the information session and approximately one hour before surgery. The goal is to determine whether visual tools provide additional benefit beyond standard counseling in reducing preoperative anxiety.

DETAILED DESCRIPTION:
This was a single-center, randomized, parallel-group study assessing the effect of different counseling tools on preoperative anxiety in patients undergoing elective bimaxillary orthognathic surgery. All participants received standardized verbal preoperative information delivered in a consistent setting. Group A received verbal information only; Group B received verbal information supplemented with an animation video; and Group C received verbal information supplemented with a 3-D anatomical skull model demonstration. Information sessions were standardized and lasted approximately 10 minutes. Anxiety was measured using the STAI (state and trait components) and a VAS at two predefined time points: baseline (before the information session) and approximately one hour before surgery. The main comparisons were changes in anxiety scores between groups to evaluate whether visual tools reduced preoperative anxiety beyond standard counseling. Data collection of anxiety assessments was performed by blinded personnel, and ethical approval and written informed consent were obtained.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years).
* Scheduled to undergo elective bimaxillary orthognathic surgery under general anesthesia.
* Able to understand the study procedures and complete the anxiety questionnaires.
* Provided written informed consent.

Exclusion Criteria:

* Current diagnosis of a major psychiatric disorder or use of anxiolytic/antidepressant medication that could affect anxiety assessment.
* Cognitive impairment or inability to complete the questionnaires.
* Emergency surgery.
* Refusal to participate or withdrawal of consent.
* Any condition judged by the investigator to interfere with participation or outcome assessment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for Anxiety (VAS-A) | From baseline (before preoperative counseling) to immediately before surgery
  Change in preoperative anxiety level measured using the Visual Analogue Scale for Anxiety (VAS-A). The scale ranges from 0 (no anxiety) to 100 (maximum anxiety).
State-Trait Anxiety Inventory | From baseline (before preoperative counseling) to immediately before surgery
  Change in state anxiety measured using the State subscale of the State-Trait Anxiety Inventory (STAI-S). The overall (total) score for STAI ranges from a minimum of 20 to a maximum of 80; STAI scores are commonly classified as 'no or low anxiety' (20-37), 'moderate anxiety' (38-44), and 'high anxiety' (45-80)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara universty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes